CLINICAL TRIAL: NCT00003259
Title: Master Protocol for Metastatic Hormone-Resistant Prostatic Carcinoma Phase II Trials Protocol 4: Vinorelbine
Brief Title: Vinorelbine in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: SAKK 08/97; SWS-SAKK-08/97; EU-97042
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vinorelbine

INTERVENTIONS:
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of vinorelbine in treating patients with metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of vinorelbine in patients with metastatic hormone-resistant prostate cancer. II. Evaluate the toxicity of vinorelbine in these patients. III. Evaluate the quality of life of these patients, and correlate quality of life with PSA response.

OUTLINE: Patients receive a 5-10 minute intravenous infusion of vinorelbine on day 1 and day 8 of a 21-day course. Patients with stabilization of their disease, partial response, or complete response, receive a maximum of 12 courses of treatment. Patients showing disease progression or severe toxic side effects discontinue treatment. Quality of life and pain are assessed prior to treatment, at days 1 and 8 of each course, and at end of the treatment. Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 14-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven metastatic stage IV prostate cancer Proven hormonal resistance Measurable or evaluable disease PSA at least 3 times upper limit of normal No leptomeningeal or brain metastases

PATIENT CHARACTERISTICS: Age: 18 to 85 Performance status: WHO 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: WBC at least 3500/mm3 OR Granulocyte count at least 2000/mm3 Hemoglobin at least 9 g/dL Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No acute severe infections No other neoplastic diseases except curatively treated basal cell or squamous cell carcinoma of the skin, or relapse free for more than 5 years after curative treatment of a neoplasm

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior cytostatic chemotherapy Endocrine therapy: At least 1 month since antiandrogens Prior hormonal therapy required Radiotherapy: No radiotherapy within the past 4 weeks No radiotherapy to the lesions used to evaluate activity of the study drug Surgery: Prior orchiectomy allowed Other: No other investigational drugs during the last month No prior therapy with cytostatic agents

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-10; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Morant, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (10):
- Switzerland (10):
  - Kantonspital Aarau, Aarau
  - Office of Walter Weber-Stadelman, Basel
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Kantonsspital - Saint Gallen, Sankt Gallen
  - Burgerspital, Solothurn, Solothurn
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich

REFERENCES:
- [Result] Morant R, Hsu Schmitz SF, Bernhard J, Thurlimann B, Borner M, Wernli M, Egli F, Forrer P, Streit A, Jacky E, Hanselmann S, Bauer J, Hering F, Schmid HP. Vinorelbine in androgen-independent metastatic prostatic carcinoma--a phase II study. Eur J Cancer. 2002 Aug;38(12):1626-32. doi: 10.1016/s0959-8049(02)00145-4. PMID 12142053